CLINICAL TRIAL: NCT00137267
Title: A Brief Community Linkage Intervention for Dually Diagnosed Individuals
Acronym: TLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIR 02-145
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Results first posted 2015-04-29 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-04

CONDITIONS: Schizophrenia; Psychotic Disorders; Substance-Related Disorders; Bipolar Disorder
Keywords: Schizophrenia / disorders w psychotic features; Substance-related disorders; Community Mental Health Services; Case Management; Health Education
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Substance-Related Disorders; Bipolar Disorder; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): This group will receive treatment as usual on Acute Psychiatry and at the Day Treatment Center along with an enhanced Time Limited Case Management community linkage intervention (TLC). Patients assigned to TLC will be offered enhanced services that begin on Acute Psychiatry and continue for a total of eight weeks through the community and Day Treatment Center transition.
  Interventions: Behavioral: Time limited case management
- Arm 2 (Active Comparator): This group will receive treatment as usual in Acute Psychiatry and at the Day Treatment Center in addition to participating in four group and one individual health education sessions (i.e., the attention control group). The length of the health education sessions (four group sessions and one individual session) will match the amount of attention provided to the treatment group. The health education sessions will cover topics such as nutrition, disease prevention, injury prevention, and healthy aging.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Time limited case management — This group will receive treatment as usual on Acute Psychiatry and at the Day Treatment Center along with an enhanced Time Limited Case Management community linkage intervention (TLC). Patients assigned to TLC will be offered enhanced services that begin on Acute Psychiatry and continue for a total of eight weeks through the community and Day Treatment Center transition.
  Other Names: TLC
  Arms: Arm 1
Behavioral: Health Education — This group will receive treatment as usual in Acute Psychiatry and at the Day Treatment Center in addition to participating in four group and one individual health education sessions (i.e., the attention control group). The length of the health education sessions (four group sessions and one individual session) will match the amount of attention provided to the treatment group. The health education sessions will cover topics such as nutrition, disease prevention, injury prevention, and healthy aging.
  Other Names: TAU+A
  Arms: Arm 2

SUMMARY:
Surveys suggest that up to 80% of veterans with a persistent mental illness have a co-occurring substance use disorder. Substance abuse among this population is problematic and often results in poor engagement in treatment and thus, frequent hospitalizations and an unstable illness course. Regarding treatment engagement, data from a VA New Jersey facility indicated that 50% of those veterans discharged from the acute psychiatric hospital unit to outpatient care did not attend their initial screening appointment and another 30% dropped out within six weeks. To assist with the transition from inpatient to outpatient care, we previously developed an eight-week augmentation intervention entitled, Time-Limited Case Management (TLC). TLC integrates evidence-based interventions of 1) Dual Recovery Therapy; 2) Critical Time Intervention Case Management along with 3) Peer Support with the goal of assisting individuals with the transition from inpatient to outpatient care.

DETAILED DESCRIPTION:
This study involved a randomized attention controlled trial of 102 individuals recruited on the inpatient psychiatry service at the New Jersey VA with a substance abuse disorder and a severe and persistent mental illness. Subjects were randomly assigned to one of two conditions: 1) treatment-as-usual in inpatient and outpatient services plus 8 weeks of Time Limited Care-Coordination (TLC), a brief linkage augmentation intervention or 2) treatment-as-usual along with 8 weeks of matched attention in the form of health education sessions (TAU+A). The data analytic plan included descriptive and advanced statistical analysis.

Objective # 1: To determine whether those in TLC have better attendance in inpatient sessions compared to those receiving Treatment-As-Usual Plus Attention (TAU+A).

Objective # 2: To determine whether those in TLC have better attendance in outpatient sessions compared to those receiving Treatment-As-Usual Plus Attention (TAU+A).

Objective # 3: To determine whether TLC, compared to Treatment-As-Usual Plus Attention (TAU+A) reduces rehospitalizations and has an effect on the use of the Emergency Room use.

Objective # 4: To determine whether TLC achieves a reduction in drug usage and related problems as compared to those receiving TAU+A.

A total of 102 veterans were randomly assigned to one of two conditions: (1) Time Limited Care-Coordination (TLC), an eight-week co-occurring disorders intervention or (2) Treatment As Usual + Matched Attention (TAU+A) control condition in the form of health education sessions. However, both groups also received treatment as usual in inpatient and outpatient settings.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients over 18 years old.
2. Patients who have a substance abuse disorder and a diagnosis of schizophrenia, schizoaffective disorder, or bipolar I disorder.
3. Patients seeking outpatient treatment for the above disorders from the VA.
4. Physically mobile
5. Agree to take public transportation if they do not have other private sources.

Exclusion Criteria:

1. Patients who only have either a mental health problem, or a substance abuse problem, but not both.
2. Patients who do not have a residence where they can stay upon discharge from the hospital.
3. Patients who are not sufficiently medically or psychiatrically stable to participate in residential or outpatient treatment. Those patients could be re-evaluated for the study once stabilized.
4. Patients exclusively engaged in methadone maintenance programs.
5. Patients who represent a serious suicide risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2005-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Smelson, PsyD, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford
Locations (2):
- United States (2):
  - Edith Nourse Rogers Memorial Veterans Hospital, Bedford, Bedford, Massachusetts
  - VA New Jersey Health Care System, East Orange, East Orange, New Jersey

REFERENCES:
- [Result] Ziedonis DM, Smelson D, Rosenthal RN, Batki SL, Green AI, Henry RJ, Montoya I, Parks J, Weiss RD. Improving the care of individuals with schizophrenia and substance use disorders: consensus recommendations. J Psychiatr Pract. 2005 Sep;11(5):315-39. doi: 10.1097/00131746-200509000-00005. PMID 16184072
- [Result] Smelson DA, Dixon L, Craig T, Remolina S, Batki SL, Niv N, Owen R. Pharmacological treatment of schizophrenia and co-occurring substance use disorders. CNS Drugs. 2008;22(11):903-16. doi: 10.2165/00023210-200822110-00002. PMID 18840032
- [Result] Sussner B, Kline A, Smelson DA, Losonczy M, Salvatore S. The role of psychosocial characteristics in irregular discharge form residentioal services for homeless veterans. Psychological Services. 2008 May 1; 5(4):341-350.
- [Result] Banerjea R, Pogach LM, Smelson D, Sambamoorthi U. Mental illness and substance use disorders among women veterans with diabetes. Womens Health Issues. 2009 Nov-Dec;19(6):446-56. doi: 10.1016/j.whi.2009.07.007. PMID 19879456
- See also: This website is intended as a source of information for anyone interested in learning more about the MISSION model (previously called TLC). — http://www.missionmodel.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Health Education: This group will receive treatment as usual in Acute Psychiatry and at the Day Treatment Center in addition to participating in four group and one individual health education sessions (i.e., the attention control group). The length of the health education sessions (four group sessions and one individual session) will match the amount of attention provided to the treatment group. The health education sessions will cover topics such as nutrition, disease prevention, injury prevention, and healthy aging.
  Health Education: This group will receive treatment as usual in Acute Psychiatry and at the Day Treatment Center in addition to participating in four group and one individual health education sessions (i.e., the attention control group). The length of the health education sessions (four group sessions and one individual session) will match the amount of attention provided to the treatment group.
Period: Overall Study
Arm/Group | Time Limited Case Management | Health Education
Started | 55 | 47
Completed | 40 | 26
Not Completed | 15 | 21
Not completed — Lost to Follow-up | 15 | 21

BASELINE CHARACTERISTICS:
Groups:
- Arm 1 - Time Limited Case Management (TLC): This group will receive treatment as usual on Acute Psychiatry and at the Day Treatment Center along with an enhanced Time Limited Case Management community linkage intervention (TLC). Patients assigned to TLC will be offered enhanced services that begin on Acute Psychiatry and continue for a total of eight weeks through the community and Day Treatment Center transition.
  Time limited case management: This group will receive treatment as usual on Acute Psychiatry and at the Day Treatment Center along with an enhanced Time Limited Case Management community linkage intervention (TLC). Patients assigned to TLC will be offered enhanced services that begin on Acute Psychiatry and continue for a total of eight weeks through the community and Day Treatment Center transition.
- Arm 2 - Health Education: This group will receive treatment as usual in Acute Psychiatry and at the Day Treatment Center in addition to participating in four group and one individual health education sessions (i.e., the attention control group). The length of the health education sessions (four group sessions and one individual session) will match the amount of attention provided to the treatment group.
  Health Education: This group will receive treatment as usual in Acute Psychiatry and at the Day Treatment Center in addition to participating in four group and one individual health education sessions (i.e., the attention control group). The length of the health education sessions (four group sessions and one individual session) will match the amount of attention provided to the treatment group. The health education sessions will cover topics such as nutrition, disease prevention, injury prevention, and healthy aging.
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Time Limited Case Management (TLC) | Arm 2 - Health Education | Total
Number analyzed (Participants) | 40 | 26 | 66
Age, Customized [Number; unit: participants]
  less than 40 years | 4 | 4 | 8
  40 - 49 years | 17 | 8 | 25
  50 and older | 19 | 14 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 38 | 26 | 64
Region of Enrollment [Number; unit: participants]
  United States | 40 | 26 | 66

OUTCOME MEASURES:

1. Primary Outcome: Treatment Engagement
Description: Number of inpatient and outpatient treatment sessions attended during the 8-week treatment period
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: number of treatment sessions attended
Groups:
- Arm 2: This group will receive treatment as usual in Acute Psychiatry and at the Day Treatment Center in addition to participating in four group and one individual health education sessions (i.e., the attention control group). The length of the health education sessions (four group sessions and one individual session) will match the amount of attention provided to the treatment group.
  Health Education: This group will receive treatment as usual in Acute Psychiatry and at the Day Treatment Center in addition to participating in four group and one individual health education sessions (i.e., the attention control group). The length of the health education sessions (four group sessions and one individual session) will match the amount of attention provided to the treatment group. The health education sessions will cover topics such as nutrition, disease prevention, injury prevention, and healthy aging.
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 40 | 26
number of treatment sessions attended
  Inpatient treatment sessions | 4.2 (3.7) | 1.4 (2.2)
  Outpatient treatment sessions | 7.2 (7.4) | 1.5 (5.2)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority or Other; p < 0.001, Chi-squared

2. Secondary Outcome: Number of Days Engaged
Description: Number of days veteran was involved with the program, from initial consent to last day of contact
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Days engaged in program
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 40 | 26
Days engaged in program | 37.3 (21.3) | 28.9 (25.1)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority or Other; p = 0.152, Chi-squared

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/26
Other Adverse Events (participants affected / at risk) | 0/40 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes